CLINICAL TRIAL: NCT01719146
Title: Computational Approach to Personalized Anemia Management
Brief Title: Prospective Observational Study of Erythropoietin-Iron Interaction in Anemia of Renal Disease
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adam Edward Gaweda, Associate Professor, University of Louisville
Other Study IDs: 12.0149; R01DK093832 (NIH)
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Anemia of End Stage Renal Disease
Keywords: Anemia; Chronic Kidney Disease; Erythropoiesis Stimulating Agents; Erythropoietin; Iron; Iron Deficiency
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Iron Deficiencies | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, serum will be extracted and frozen for further analysis. Serum will be retained for up to 60 days.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- UofL Subjects: Subjects undergoing Specimen Collection at University Kidney Center, University of Louisville, Louisville, KY
  Interventions: Other: Specimen collection
- Duke Subjects: Subjects undergoing Specimen Collection at Duke University, Durham, NC
  Interventions: Other: Specimen collection
- WNERTA Subjects: Subject undergoing Specimen Collection at Western New England Renal and Transplant Associates, Springfield, MA
  Interventions: Other: Specimen collection

INTERVENTIONS:
Other: Specimen collection — At the beginning of each midweek hemodialysis session, a blood specimen (4 mL) will be drawn from the study subject. Out of this specimen a 1 mL serum sample will be frozen and stored. A 3 mL blood sample will be shipped overnight to WNERTA for laboratory testing.

SUMMARY:
The purpose of this study is to prospectively collect data on doses of Erythropoietic Stimulating Agents (ESA) and Intravenous Iron, and the markers of erythropoietic activity and iron status. These data will be used to derive mathematical models which will subsequently guide dosing of both agents, such that a desired therapeutic outcome is achieved in every patient, while minimizing patient exposure to both agents.

DETAILED DESCRIPTION:
Data will be collected from 120 subjects undergoing hemodialysis treatment at 3 clinical sites across United States (40 per site).5.5 mL blood specimen will be drawn during midweek treatment (Wed/Thu) to measure:

Hemoglobin Concentration Hematocrit Red Blood Cell Count Platelet Count Reticulocyte Percentage Reticulocyte Hemoglobin Mean Cellular Hemoglobin Mean Cellular Hemoglobin Concentration Mean Cell Volume Red Cell Volume Distribution Width Mean Platelet Volume Serum Iron Serum Ferritin Transferrin Saturation Hepcidin Soluble Transferrin Receptor

Weekly ESA and Iron dose delivered will also be recorded.

From these data:

1. a mathematical model will be established to find biomarkers most descriptive with respect to erythropoiesis-iron synergy,
2. a mathematical model will be established to correlate iron dose with iron markers.

ELIGIBILITY:
Inclusion Criteria:

* receiving or expected to receive ESA

Exclusion Criteria:

* life expectancy less than 12 months
* frequent (once or more per month w/in last 6 months) uncontrolled blood loss
* frequent (once or more per month w/in last 6 months) hospitalization
* frequent (once or more per month w/in last 6 months) access complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End Stage Renal Disease Patients undergoing hemodialysis treatments at:
  1. University Kidney Center, Louisville, KY
  2. Duke University, Durham, NC
  3. WNERTA, Springfield, MA
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2013-01; Primary Completion 2021-06-05 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Concentration (g/dL) | 52 weeks
  Weekly Hemoglobin Concentration

OTHER OUTCOMES:
Transferrin Saturation (%) | 52 weeks
  Weekly Transferrin Saturation
Serum Ferritin (ng/mL) | 52 weeks
  Weekly Serum Ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Adam E Gaweda, Ph.D., Principal Investigator — University of Louisville
Locations (3):
- United States (3):
  - University of Louisville, University Kidney Center, Louisville, Kentucky
  - Western New England Renal and Transplant Associates, Springfield, Massachusetts
  - Duke University, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided